CLINICAL TRIAL: NCT00197145
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter, Parallel Group Study to Compare the Efficacy and Safety of GW873140 400mg BID in Combination With a Ritonavir-containing Optimized Background Therapy (OBT) Regimen Versus Placebo Plus OBT Over 48 Weeks.
Brief Title: Study Of Chemokine Coreceptor 5 (CCR5) Antagonist GW873140 In R5-Tropic Treatment-Experienced HIV-Infected Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: CCR102709
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus I
Keywords: HIV-1 GW873140 CCR5 antagonist experienced
MeSH Terms: conditions — Infections | interventions — aplaviroc

ARMS (1):
- GW873140 (Experimental)
  Interventions: Drug: GW873140

INTERVENTIONS:
Drug: GW873140 — 400 mg twice daily

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the CCR5 antagonist GW873140 or placebo in combination with an optimized background regimen in treatment-experienced HIV-infected subjects with R5-tropic virus

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected.
* Screening viral load at least 5000copies/mL.
* R5-tropic only virus at screening.
* Total prior antiretroviral experience of at least 3 months and documented resistance to at least one drug in each of the following classes: nucleoside reverse transcriptase inhibitors (NRTI), non-nucleoside reverse transcriptase inhibitors (NNRTI), and protease inhibitors (PI).
* Stable antiretroviral regimen (or no antiretroviral treatment) for at least 4 weeks before screening.
* Able to receive a ritonavir-boosted protease inhibitor during treatment studies.
* Women of childbearing potential must use specific forms of contraception.

Exclusion criteria:

* Acute laboratory abnormalities.
* History of pancreatitis or hepatitis, hepatitis B or hepatitis C coinfection, or any chronic liver disease. Screening liver function tests will be used to determine eligibility.
* R5/X4-tropic, X4-tropic only, or non-phenotypeable virus at screening.
* Changes to antiretroviral therapy from 4 weeks prior to screening until Day 1 of treatment study.
* Pregnancy or breastfeeding women.
* Recent participation in an experimental drug trial.
* Prior use of a CCR5 or CXCR4 antagonist.
* Significant ECG abnormalities or significant history of active pancreatitis, hepatitis, opportunistic infections, malabsorption disorders, cancer, or severe illness.
* Current use of certain medications may exclude participation in this study.
* Additional qualifying criteria and laboratory test requirements to be assessed by study physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-07-21 (Actual); Primary Completion 2007-09-11 (Actual); Study Completion 2007-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (49):
- United States (46):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Laguna Beach, California
  - GSK Investigational Site, Long Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Glastonbury, Connecticut
  - GSK Investigational Site, Norwalk, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Fort Myers, Florida
  - GSK Investigational Site, Key West, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Oakland Park, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Plantation, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Portland, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Hillsborough, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Mount Vernon, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Akron, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Annandale, Virginia
  - GSK Investigational Site, Hampton, Virginia
  - GSK Investigational Site, Lynchburg, Virginia
  - GSK Investigational Site, Spokane, Washington
- GSK Investigational Site, Toronto, Ontario, Canada
- Puerto Rico (2):
  - GSK Investigational Site, Ponce
  - GSK Investigational Site, San Juan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was planned on 406 male or female participants infected with Human immunodeficiency type 1 (HIV-1) virus, aged 18 years or older, across 15 centres in the United States and at 1 site in Canada from 21 July 2005 to 11 September 2007. Study was early terminated prior to the completion of enrollment.
Pre-assignment Details: A total of 24 participants comprised All Randomized Subject Population who were randomized in a ratio of 1:1 to GW873140 (aplaviroc [APL])+optimized background therapy (OBT) and placebo+OBT. Intent-to Treat (ITT) Population was n=24, used for all analysis.
Groups:
- APL + OBT: Participants were administered APL tablets orally as 400 milligram (mg) twice daily (BID) for 48 Weeks. Each dose was to be given with food. The OBT regimen was chosen by the investigator prior to randomization, based on the participant's prior treatment history, screening genotypic and phenotypic resistance testing results, and any prior resistance testing results if available. The drugs in the OBT regimen was chosen from the locally available ART and consisted between three and six drugs, one of which was ritonavir (RTV)- boosted protease inhibitor (PI). Low-dose RTV did not count as one of the OBT regimen drugs and RTV doses of >400 mg/day were not permitted. Fixed dose combination tablets (FDC) was counted according to the number of compounds making up the FDC (e.g., combivir counted as two drugs [lamivudine and zidovudine], trizivir counted as three drugs, etc.). Kaletra (lopinavir [LPV]/RTV) was counted as one drug.
- Placebo + OBT: Participants were administered matching placebo to APL tablets orally as 400 mg BID for 48 Weeks. Each dose was to be given with food. The OBT regimen was chosen by the investigator prior to randomization, based on the participant's prior treatment history, screening genotypic and phenotypic resistance testing results, and any prior resistance testing results if available. The drugs in the OBT regimen was chosen from the locally available ART and consisted between three and six drugs, one of which was ritonavir (RTV)- boosted protease inhibitor (PI). Low-dose RTV did not count as one of the OBT regimen drugs and RTV doses of >400 mg/day were not permitted. Fixed dose combination tablets (FDC) was counted according to the number of compounds making up the FDC (e.g., combivir counted as two drugs [lamivudine and zidovudine], trizivir counted as three drugs, etc.). Kaletra (lopinavir [LPV]/RTV) was counted as one drug.
Period: Period 1: Randomized Treatment Phase
Arm/Group | APL + OBT | Placebo + OBT
Started | 13 | 11
Completed | 0 | 0
Not Completed | 13 | 11
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Sponsor terminated study | 10 | 8
Not completed — Other | 2 | 2
Period: Period 2 : Open Label Phase
Arm/Group | APL + OBT | Placebo + OBT
Started | 10 | 0
Completed | 0 | 0
Not Completed | 10 | 0
Not completed — Insufficient viral load response | 1 | 0
Not completed — Protocol defined virological failure | 3 | 0
Not completed — Availability of alternative ART | 2 | 0
Not completed — Were ongoing till data freeze | 3 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- APL + OBT: Participants were administered APL tablets orally as 400 mg BID for 48 Weeks. Each dose was to be given with food. The OBT regimen was chosen by the investigator prior to randomization, based on the participant's prior treatment history, screening genotypic and phenotypic resistance testing results, and any prior resistance testing results if available. The drugs in the OBT regimen was chosen from the locally available ART and consisted between three and six drugs, one of which was RTV-boosted PI. Low-dose RTV did not count as one of the OBT regimen drugs and RTV doses of >400 mg/day were not permitted. FDC was counted according to the number of compounds making up the FDC (e.g., combivir counted as two drugs [lamivudine and zidovudine], trizivir counted as three drugs, etc.). Kaletra (LPV/RTV) was counted as one drug.
- Placebo + OBT: Participants were administered matching placebo to APL tablets orally as 400 mg BID for 48 Weeks. Each dose was to be given with food. The OBT regimen was chosen by the investigator prior to randomization, based on the participant's prior treatment history, screening genotypic and phenotypic resistance testing results, and any prior resistance testing results if available. The drugs in the OBT regimen was chosen from the locally available ART and consisted between three and six drugs, one of which was RTV-boosted PI. Low-dose RTV did not count as one of the OBT regimen drugs and RTV doses of >400 mg/day were not permitted. FDC was counted according to the number of compounds making up the FDC (e.g., combivir counted as two drugs [lamivudine and zidovudine], trizivir counted as three drugs, etc.). Kaletra (LPV/RTV) was counted as one drug.
- Total: Total of all reporting groups
Arm/Group | APL + OBT | Placebo + OBT | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.8 (7.03) | 44.5 (5.68) | 45.8 (6.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 11 | 9 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Plasma HIV-1 RNA <400 Copies Per Milliliter (Copies /mL) at Week 24 and 48
Description: Assessment for plasma HIV-1 RNA was done at Week 24 and also planned at Week 48 by polymerase chain reaction (PCR) analysis. Data is reported for number of participants with plasma HIV-1 RNA <400 copies/mL at Week 24. Data was not collected for Week 48 due to early termination of the study.
Time Frame: Week 24
Population: Intent to Treat (ITT) Population comprised of all participants randomized with evidence of receiving at least one dose of study medication. The analysis was an observed analysis and only participants with data available at the indicated timepoints were included.
Measure: Count of Participants; unit: Participants
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 7 | 0
Participants | 5 | 0

2. Primary Outcome: Average Area Under the Curve Minus Baseline (AAUCMB) of Plasma HIV-1 RNA Through the Entire Study Period
Description: The area under the plasma HIV-1 RNA curve (AUC) was computed using the trapezoidal rule for all assessments (scheduled and unscheduled) at their actual time points. Baseline was defined as the mean of the Baseline (Day 1) and pre-treatment visit values. Participants without a Baseline assessment was removed from the analysis. The AAUCMB was computed by the AUC divided by the duration of the profile (i.e., the number of days on randomized therapy) minus the Baseline measurement. Data is reported up to Week 40 only due to early termination of the study.
Time Frame: Up to Week 40
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Log10 copies/mL
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 11 | 7
Log10 copies/mL | -2.03 (0.990) | -1.14 (0.766)

3. Primary Outcome: Number of Participants With >= 1.0 log10 Copies/mL Decrease in Plasma HIV-1 RNA From Baseline Over Time
Description: The plasma HIV-1 RNA polymerase chain reaction (PCR) assessments were planned at pre-Baseline (between 1 and 14 days prior to Day 1), up to Week 12 Follow- up of the Randomized Phase, up to Week 12 Follow-up of the Open Labeled Non-Randomized phase and every 6 months Follow-up of off study drug/on study phase, however the study was early terminated at Week 40. Baseline was defined as the mean of the Baseline (Day 1) and pre-treatment visit values.
Time Frame: Day 1 up to Week 12 Follow-up of the Randomized Treatment phase, up to Week 12 Follow-up of the Open Labeled Non-Randomized phase and every 6 months Follow-up of off study drug/on study phase
Population: ITT Population. Data were not collected for this outcome measure due to early termination of the study.
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants With Plasma HIV-1 RNA <50 Copies/mL at Week 24 and 48
Description: Assessment for plasma HIV-1 RNA was done at Week 24 and also planned at Week 48 by PCR analysis. Data is reported for number of participants with plasma HIV-1 RNA <50 copies/mL at Week 24. Data was not collected for Week 48 due to early termination of the study.
Time Frame: Week 24
Population: ITT Population. The analysis was an observed analysis and only participants with data available at the indicated timepoints were included.
Measure: Count of Participants; unit: Participants
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 7 | 0
Participants | 5 | 0

5. Secondary Outcome: Number of Participants With Any Adverse Event (AE), Serious Adverse Event (SAE), Death, Drug-related AE and AE Leading to Treatment Discontinuation
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, hypersensitivity reaction to abacavir. AEs were classified as potentially drug-related, based on the investigator's judgment.
Time Frame: Up to Follow-up (Week 52)
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Participants
  Any AE | 11 | 5
  Any SAE | 0 | 0
  Any Death | 0 | 0
  Drug-related AE | 7 | 2
  Any AE Leading to Treatment Discontinuation | 0 | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Laboratory Abnormalities for Chemistry Data at Any Visit Post-Baseline
Description: The participants with treatment emergent toxicities of laboratory abnormalities for chemistry data is reported . Participants with toxicities were categorized according to the division of AIDS (DAIDS) toxicity grading scale. Scale ranges from grade 1(mild)=symptoms causing no or minimal interference with usual social & functional activities, grade 2 (moderate)=symptoms causing greater than minimal interference with usual social & functional activities, grade 3 (severe)=symptoms causing inability to perform usual social & functional activities and grade 4 (potentially life threatening)=symptoms causing inability to perform basic self-care functions or medical or operative intervention indicated to prevent permanent impairment, persistent disability, or death. Scale ranges from 1-4, where higher grade reflects greater severity of symptoms. Baseline was defined as assessments done at Day 1. Only those parameters for which at least one value of toxicity grade was reported are summarized.
Time Frame: Up to Week 40
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Participants
  Alanine Amino Transferase (ALT), Grade 1 | 0 | 1
  ALT, Grade 2 | 1 | 0
  Albumin, Grade 2 | 1 | 0
  Alkaline Phosphatase (ALP), Grade 1 | 2 | 3
  Aspartate Amino Transferase (AST), Grade 1 | 1 | 2
  AST, Grade 2 | 1 | 0
  Carbon Dioxide content/Bicarbonate (CO2), Grade 1 | 2 | 3
  Cholesterol, Grade 1 | 0 | 1
  Cholesterol, Grade 2 | 1 | 0
  Creatine Kinase (CK), Grade 1 | 0 | 1
  CK, Grade 2 | 1 | 0
  CK, Grade 3 | 2 | 0
  Creatinine, Grade 1 | 1 | 2
  Glucose, Grade 1 | 3 | 3
  Glucose, Grade 2 | 3 | 2
  Glucose, Grade 3 | 1 | 0
  Low Density lipoprotein (LDL) Cholesterol, Grade 2 | 1 | 0
  Lipase, Grade 1 | 3 | 0
  Lipase, Grade 2 | 1 | 0
  Potassium, Grade 4 | 0 | 1
  Sodium, Grade 1 | 3 | 2
  Total Bilirubin, Grade 1 | 0 | 1
  Total Bilirubin, Grade 2 | 1 | 0
  Total Bilirubin, Grade 4 | 1 | 0
  Triglycerides, Grade 2 | 0 | 2
  Triglycerides, Grade 3 | 1 | 0

7. Secondary Outcome: Change From Baseline in Chemistry Parameters of ALT, ALP, AST and CK During the Randomized Treatment Phase
Description: Assessment was performed at Day 1, Week 12 and Week 24. Baseline was defined as the assessments done at Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Week 12 and 24) values.
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: International unit per liter (IU/L)
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
International unit per liter (IU/L)
  ALT, Week 12: number analyzed (Participants) | 13 | 4
  ALT, Week 12 | -7.231 (28.5048) | 9.250 (18.8569)
  ALT, Week 24: number analyzed (Participants) | 7 | 0
  ALT, Week 24 | -5.429 (19.4324) |
  ALP, Week 12: number analyzed (Participants) | 13 | 4
  ALP, Week 12 | -7.154 (24.1069) | 25.750 (18.9275)
  ALP, Week 24: number analyzed (Participants) | 7 | 0
  ALP, Week 24 | -3.571 (19.4753) |
  AST, Week 12: number analyzed (Participants) | 13 | 4
  AST, Week 12 | -4.231 (15.9330) | 4.750 (8.4212)
  AST, Week 24: number analyzed (Participants) | 7 | 0
  AST, Week 24 | -3.857 (13.5699) |
  CK, Week 12: number analyzed (Participants) | 13 | 4
  CK, Week 12 | -3.462 (185.5095) | 37.250 (78.9910)
  CK, Week 24: number analyzed (Participants) | 7 | 0
  CK, Week 24 | 102.714 (553.4250) |

8. Secondary Outcome: Change From Baseline in Chemistry Parameters of CO2 Content/Bicarbonate, Chloride, Cholesterol, Glucose, High DL Cholesterol, LDL Cholesterol, Triglycerides, Potassium, Urea and Sodium During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimole (MMOL)/L
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Millimole (MMOL)/L
  CO2 content/bicarbonate, Week 12: number analyzed (Participants) | 13 | 4
  CO2 content/bicarbonate, Week 12 | 0.154 (2.5445) | -1.250 (4.1932)
  CO2 content/bicarbonate, Week 24: number analyzed (Participants) | 7 | 0
  CO2 content/bicarbonate, Week 24 | 2.429 (3.6450) |
  Chloride, Week 12: number analyzed (Participants) | 13 | 4
  Chloride, Week 12 | 0.462 (3.4306) | -2.500 (2.6458)
  Chloride, Week 24: number analyzed (Participants) | 7 | 0
  Chloride, Week 24 | 0.857 (2.7946) |
  Cholesterol, Week 12: number analyzed (Participants) | 7 | 1
  Cholesterol, Week 12 | -0.200 (0.7095) | -0.700 (NA) — SD was not generated as only 1 participant was assessed during this time point.
  Cholesterol, Week 24: number analyzed (Participants) | 7 | 0
  Cholesterol, Week 24 | -0.539 (0.8367) |
  Glucose, Week 12: number analyzed (Participants) | 13 | 4
  Glucose, Week 12 | 0.415 (3.2246) | 1.150 (1.3964)
  Glucose, Week 24: number analyzed (Participants) | 7 | 0
  Glucose, Week 24 | -0.357 (1.8063) |
  HDL, Week 12: number analyzed (Participants) | 7 | 1
  HDL, Week 12 | -0.036 (0.2340) | -0.100 (NA) — SD was not generated as only 1 participant was assessed during this time point.
  HDL, Week 24: number analyzed (Participants) | 7 | 0
  HDL, Week 24 | 0.026 (0.2028) |
  LDL, Week 12: number analyzed (Participants) | 6 | 1
  LDL, Week 12 | -0.552 (0.5635) | -0.500 (NA) — SD was not generated as only 1 participant was assessed during this time point.
  LDL, Week 24: number analyzed (Participants) | 7 | 0
  LDL, Week 24 | -0.597 (0.6607) |
  Potassium, Week 12: number analyzed (Participants) | 13 | 4
  Potassium, Week 12 | 0.038 (0.3906) | -0.225 (0.3304)
  Potassium, Week 24: number analyzed (Participants) | 7 | 0
  Potassium, Week 24 | -0.114 (0.1952) |
  Sodium, Week 12: number analyzed (Participants) | 13 | 4
  Sodium, Week 12 | -0.846 (1.5730) | -2.500 (3.6968)
  Sodium, Week 24: number analyzed (Participants) | 7 | 0
  Sodium, Week 24 | 0.714 (1.9760) |
  Triglycerides, Week 12: number analyzed (Participants) | 7 | 1
  Triglycerides, Week 12 | 1.194 (1.3095) | -0.240 (NA) — SD was not generated as only 1 participant was assessed during this time point.
  Triglycerides, Week 24: number analyzed (Participants) | 7 | 0
  Triglycerides, Week 24 | 0.071 (0.7076) |
  Urea, Week 12 | -0.162 (2.3835) | 0.375 (2.9545)
  Urea, Week 24: number analyzed (Participants) | 7 | 0
  Urea, Week 24 | -0.343 (2.3572) |

9. Secondary Outcome: Change From Baseline in Chemistry Parameter of Creatinine and Total Bilirubin During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromole (UMOL)/L
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Micromole (UMOL)/L
  Creatinine, Week 12: number analyzed (Participants) | 13 | 4
  Creatinine, Week 12 | -1.385 (11.3397) | 13.000 (11.1056)
  Creatinine, Week 24: number analyzed (Participants) | 7 | 0
  Creatinine, Week 24 | -2.714 (12.7504) |
  Total Bilirubin, Week 12: number analyzed (Participants) | 13 | 4
  Total Bilirubin, Week 12 | 0.769 (18.8244) | -0.500 (6.8069)
  Total Bilirubin, Week 24: number analyzed (Participants) | 7 | 0
  Total Bilirubin, Week 24 | 8.286 (31.0790) |

10. Secondary Outcome: Change From Baseline in Chemistry Parameter of Albumin During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed
Measure: Mean (Standard Deviation); unit: Gram (g)/L
Groups:
- APL + OBT; Placebo + OBT: Participants were administered matching placebo to APL tablets orally as 400 mg BID for 48 Weeks. Each dose was to be given with food. The OBT regimen was chosen by the investigator prior to randomization, based on the participant's prior treatment history, screening genotypic and phenotypic resistance testing results, and any prior resistance testing results if available. The drugs in the OBT regimen was chosen from the locally available ART and consisted between three and six drugs, one of which was RTV-boosted PI. Low-dose RTV did not count as one of the OBT regimen drugs and RTV doses of >400 mg/day were not permitted. FDC was counted according to the number of compounds making up the FDC (e.g., combivir counted as two drugs [lamivudine and zidovudine], trizivir counted as three drugs, etc.). Kaletra (LPV/RTV) was counted as one drug.
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Gram (g)/L
  Week 12: number analyzed (Participants) | 13 | 4
  Week 12 | 1.385 (2.6627) | 3.750 (2.5000)
  Week 24: number analyzed (Participants) | 7 | 0
  Week 24 | 2.000 (3.5590) |

11. Secondary Outcome: Change From Baseline in Chemistry Parameter of Lipase During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
U/L
  Week 12: number analyzed (Participants) | 11 | 2
  Week 12 | 6.636 (8.4531) | 0.000 (4.2426)
  Week 24: number analyzed (Participants) | 7 | 0
  Week 24 | 12.571 (20.3867) |

12. Secondary Outcome: Change From Baseline in Haematology Parameters of Basophils, Eosinophils, Lymphocytes, Monocytes, Platelet Count, Total Neutrophils, White Blood Cell (WBC) Count During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells (GI)/L
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Giga cells (GI)/L
  Basophils, Week 12: number analyzed (Participants) | 13 | 2
  Basophils, Week 12 | -0.003 (0.0085) | -0.005 (0.0212)
  Basophils, Week 24: number analyzed (Participants) | 7 | 0
  Basophils, Week 24 | -0.000 (0.0153) |
  Eosinophils, Week 12: number analyzed (Participants) | 13 | 2
  Eosinophils, Week 12 | -0.027 (0.1013) | 0.090 (0.1697)
  Eosinophils, Week 24: number analyzed (Participants) | 7 | 0
  Eosinophils, Week 24 | -0.010 (0.0876) |
  Lymphocytes, Week 12: number analyzed (Participants) | 13 | 2
  Lymphocytes, Week 12 | 0.573 (0.4762) | 0.050 (0.2970)
  Lymphocytes, Week 24: number analyzed (Participants) | 7 | 0
  Lymphocytes, Week 24 | 0.373 (0.7915) |
  Monocytes, Week 12: number analyzed (Participants) | 13 | 2
  Monocytes, Week 12 | 0.041 (0.1398) | -0.095 (0.2758)
  Monocytes, Week 24: number analyzed (Participants) | 7 | 0
  Monocytes, Week 24 | 0.079 (0.0756) |
  Platelet Count, Week 12: number analyzed (Participants) | 13 | 2
  Platelet Count, Week 12 | 47.846 (38.5202) | -3.500 (33.2340)
  Platelet Count, Week 24: number analyzed (Participants) | 7 | 0
  Platelet Count, Week 24 | 70.143 (51.2199) |
  Total Neutrophils, Week 12: number analyzed (Participants) | 13 | 2
  Total Neutrophils, Week 12 | 0.963 (1.0130) | -0.935 (0.3889)
  Total Neutrophils, Week 24: number analyzed (Participants) | 7 | 0
  Total Neutrophils, Week 24 | 0.861 (0.9786) |
  WBC Count, Week 12: number analyzed (Participants) | 13 | 2
  WBC Count, Week 12 | 1.546 (1.1125) | -0.900 (1.1314)
  WBC Count, Week 24: number analyzed (Participants) | 7 | 0
  WBC Count, Week 24 | 1.300 (1.1015) |

13. Secondary Outcome: Change From Baseline in Haematology Parameter of Mean Corpuscle Volume (MCV) During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtoliter (FL)
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Femtoliter (FL)
  Week 12: number analyzed (Participants) | 13 | 2
  Week 12 | -3.000 (7.7567) | -1.500 (4.9497)
  Week 24: number analyzed (Participants) | 7 | 0
  Week 24 | -3.429 (9.5019) |

14. Secondary Outcome: Change From Baseline in Haematology Parameter of Hematocrit During the Randomized Treatment Phase.
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Percentage of red blood cells
  Week 12: number analyzed (Participants) | 13 | 2
  Week 12 | 0.010 (0.0354) | 0.026 (0.0099)
  Week 24: number analyzed (Participants) | 7 | 0
  Week 24 | -0.022 (0.0344) |

15. Secondary Outcome: Change From Baseline in Haematology Parameter of Hemoglobin During the Randomized Treatment Phase
Description: as for outcome 7
Time Frame: Baseline (Day 1), Week 12 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
g/L
  Week 12: number analyzed (Participants) | 13 | 2
  Week 12 | 4.923 (9.9621) | 6.500 (4.9497)
  Week 24: number analyzed (Participants) | 7 | 0
  Week 24 | -4.000 (10.2144) |

16. Secondary Outcome: Change From Baseline in Electrocardiograph (ECG) Parameter of Heart Rate (HR) During the Randomized Treatment Phase
Description: 12-lead ECG assessments were obtained at Day 1 (triplicate measurements), Week 4 and Week 24. The assessments were done using an ECG machine that automatically calculated the heart rate. Baseline was defined as the mean of the triplicate assessment done at Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Week 4 and 24) values.
Time Frame: Baseline (Day 1), Week 4 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (Bpm)
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Beats per minute (Bpm)
  Week 4: number analyzed (Participants) | 11 | 10
  Week 4 | 5.6 (12.74) | 4.3 (11.54)
  Week 24: number analyzed (Participants) | 6 | 0
  Week 24 | -3.9 (8.11) |

17. Secondary Outcome: Change From Baseline in ECG Parameter of RR Interval, Uncorrected QT Interval, QTc Interval (Fridericia), QTc Interval (Bazette), PR Interval and QRS Duration During the Randomized Treatment Phase
Description: 12-lead ECG assessments were obtained at Day 1 (triplicate measurements), Week 4 and Week 24. The assessments were done using an ECG machine that automatically measured RR, PR, QRS, uncorrected QT, QTc (Bazette) and QTc (Fridericia) intervals. Baseline was defined as the mean of the triplicate assessment done at Day 1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Week 4 and Week 24) values.
Time Frame: Baseline (Day 1), Week 4 and Week 24
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millisecond (msec)
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Millisecond (msec)
  RR Interval, Week 4: number analyzed (Participants) | 11 | 10
  RR Interval, Week 4 | -69.8 (112.21) | -52.1 (128.19)
  RR Interval, Week 24: number analyzed (Participants) | 6 | 0
  RR Interval, Week 24 | 52.2 (73.16) |
  Uncorrected QT Interval, Week 4: number analyzed (Participants) | 11 | 10
  Uncorrected QT Interval, Week 4 | -18.3 (30.87) | 1.2 (28.81)
  Uncorrected QT Interval, Week 24: number analyzed (Participants) | 6 | 0
  Uncorrected QT Interval, Week 24 | 2.5 (12.49) |
  QTc Interval (Fridericia), Week 4: number analyzed (Participants) | 11 | 10
  QTc Interval (Fridericia), Week 4 | -9.3 (26.05) | 10.2 (14.06)
  QTc Interval (Fridericia), Week 24: number analyzed (Participants) | 6 | 0
  QTc Interval (Fridericia), Week 24 | -5.2 (13.00) |
  QTc Interval (Bazette), Week 4: number analyzed (Participants) | 11 | 10
  QTc Interval (Bazette), Week 4 | -4.5 (27.68) | 15.4 (14.64)
  QTc Interval (Bazette), Week 24: number analyzed (Participants) | 6 | 0
  QTc Interval (Bazette), Week 24 | -8.8 (17.47) |
  PR Interval, Week 4: number analyzed (Participants) | 11 | 10
  PR Interval, Week 4 | -8.2 (16.24) | 0.2 (15.98)
  PR Interval, Week 24: number analyzed (Participants) | 6 | 0
  PR Interval, Week 24 | 2.5 (10.07) |
  QRS Duration, Week 4: number analyzed (Participants) | 11 | 10
  QRS Duration, Week 4 | 3.2 (7.08) | 0.4 (7.13)
  QRS Duration, Week 24: number analyzed (Participants) | 6 | 0
  QRS Duration, Week 24 | -1.3 (7.68) |

18. Secondary Outcome: Change From Baseline in Cluster of Differentiation 4 (CD4) Cell Counts During the Randomized Treatment Phase
Description: The CD4 cell count is an indication of the strength of the immune system. The assessment of CD4 cell count was done by flow cytometry. Baseline was defined as the mean of the Baseline (Day 1) and pre-treatment visit values. Change from Baseline was calculated by subtracting the Baseline value from the individual post-Baseline (Week 12, 24 and 40) values.
Time Frame: Baseline (Day 1), Week 12, Week 24 and Week 40
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Cells/Cubic millimeter (mm^3)
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Cells/Cubic millimeter (mm^3)
  Week 12: number analyzed (Participants) | 11 | 2
  Week 12 | 55.909 (53.8878) | 80.500 (177.4838)
  Week 24: number analyzed (Participants) | 7 | 0
  Week 24 | 27.000 (104.1441) |
  Week 40: number analyzed (Participants) | 3 | 0
  Week 40 | 153.000 (57.6888) |

19. Secondary Outcome: Time to Centres for Disease Control and Prevention (CDC) Class C Acquired Immune Deficiency Syndrome (AIDS)-Defining Event or Death
Description: The time to CDC class C AIDS-defining event or death was planned to be assessed as per the CDC 1993 revised classification system for HIV infection and expanded surveillance case definition for AIDS among adolescents and adults. The CDC classifies HIV infection as Category A (participants with asymptomatic HIV infection, acute HIV infection with accompanying illness, or persistent generalized lymphadenopathy), Category B (participants with symptomatic non-AIDS condition, i.e., conditions that are attributed to HIV infection or are indicative of a defect in cell-mediated immunity; or conditions are considered by physicians to have a clinical course or to require management that is complicated by HIV infection), and Category C (includes AIDS indicator conditions as defined by diagnostic or presumptive measures).
Time Frame: Up to Week 12 Follow-up of the Randomized phase, up to Week 12 Follow-up of the Open Labeled Non-Randomized phase and every 6 months Follow-up of off study drug/on study phase
Population: ITT Population. Data were not collected for this outcome measure due to early termination of the study.
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 0 | 0

20. Secondary Outcome: Number of Participants With Development of Antiretroviral Resistance to GW873140 400 mg BID and Other Antiretroviral Drugs
Description: Assessment for the development of antiretroviral resistance was performed at each visit up to Follow-up. The genotypic analysis of viral resistance associated mutations was done using protease and reverse transcriptase enzymes. The number of participants with treatment emergent changes in reverse transcriptase and protease genotypic mutations were reported.
Time Frame: Up to Follow-up (Week 52)
Population: Virologic Failure Population was defined as the number of participants with protocol defined virologic failure criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 6 | 3
Participants | 2 | 1

21. Secondary Outcome: Number of Participants With 50% Inhibitory Concentration (IC50) Fold Resistance at Baseline
Description: The IC50 is a measure of the effectiveness of a substance in inhibiting a specific biological or biochemical function. IC50 was collected for abacavir (ABC), atazanavir (ATV), delavirdine (DLV), didanosine (DDI), efavirenz (EFV), emtricitabine, enfuvirtide , fosamprenavir (AMP), GW873140 (APL), indinavir (IDV), indinavir rooted with ritonavir (IDV/r), lamivudine, lopinavir rooted with ritonavir (LPV/r), nelfinavir (NFV), nevirapine (NVP), ritonavir (RTV), saquinavir (SQV), stavudine, tenofovir (TFV), tipranavir rooted with ritonavir (TPV/r), zidovudine (ZDV). Data is categorized for number of participants with each IC50 concentration of the individual drugs at Baseline (Day 1).
Time Frame: Baseline (Day 1)
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 13 | 11
Participants
  ABC < 4.5 | 0 | 4
  ABC >= 4.5 | 13 | 7
  ATV < 2.3 | 1 | 3
  ATV >= 2.3 | 12 | 8
  ATV/r < 5.2 | 1 | 5
  ATV/r >= 5.2 | 12 | 6
  DLV < 2.5 | 3 | 4
  DLV >= 2.5 | 10 | 7
  DDI < 1.3 | 0 | 5
  DDI >= 1.3 | 13 | 6
  EFV < 2.5 | 2 | 2
  EFV >= 2.5 | 11 | 9
  Emtricitabine < 3.5 | 0 | 3
  Emtricitabine >= 3.5 | 13 | 8
  Enfuvirtide < 2.5 | 2 | 7
  Enfuvirtide >= 2.5 | 9 | 2
  AMP < 2 | 1 | 4
  AMP >= 2 | 12 | 7
  APL < 2.5 | 12 | 9
  APL >= 2.5 | 0 | 0
  IDV < 2.1 | 1 | 3
  IDV >= 2.1 | 12 | 8
  IDV/r < 10 | 2 | 7
  IDV/r >= 10 | 11 | 4
  Lamivudine < 3.5 | 0 | 4
  Lamivudine >= 3.5 | 13 | 7
  LPV/r < 10 | 3 | 6
  LPV/r >= 10 | 10 | 5
  NFV < 2.5 | 1 | 3
  NFV >= 2.5 | 12 | 8
  NVP < 2.5 | 1 | 2
  NVP >= 2.5 | 12 | 9
  RTV < 2.5 | 1 | 3
  RTV >= 2.5 | 12 | 8
  SQV < 1.7 | 1 | 3
  SQV >= 1.7 | 12 | 8
  Stavudine < 1.7 | 1 | 5
  Stavudine >= 1.7 | 12 | 6
  TFV < 1.4 | 4 | 4
  TFV >= 1.4 | 9 | 7
  TPV/r < 4 | 7 | 7
  TPV/r >= 4 | 6 | 3
  ZDV < 1.9 | 1 | 3
  ZDV >= 1.9 | 12 | 8

22. Secondary Outcome: Plasma GW873140 400 mg BID Pharmacokinetic (PK) Parameter of Area Under the Plasma Concentration-time Curve During One Dosing Interval of Length (Tau) (AUC [0-tau]) During the Randomized Treatment Phase
Description: AUC (0- tau) GW873140 was defined as the area under the plasma concentration-time curve from time 0 to tau. Blood samples for evaluation of GW873140 plasma PK was planned to be collected from all participants at Week 4, 12, and 24. Intensive PK sampling was planned to be conducted with the enrolled participants. All participants who were not part of the intensive PK group was planned to be part of the limited PK sample group. Participants were supposed to complete a diary card with the date and time of investigational product administration of the last dose prior to clinic visits on Weeks 4, 12, and 24. It was determined using the linear trapezoidal rule for increasing concentrations and the logarithmic trapezoidal rule for decreasing concentrations.
Time Frame: Week 4 (pre-dose [0 hour], 1, 2, 3, 4, 6, 8, 10 hour post-evening dose), Week 12 (pre-dose [0 hour] and 2-4 hour post-morning dose) and Week 24 (pre-dose and 2-4 hour post-morning dose)
Population: The PK Population was defined as all participants who received GW873140 and underwent plasma PK sampling during the study. Participants for whom plasma a PK sample was obtained and assayed were planned to be included in analyses of the PK population. Data were not collected for this outcome measure due to early termination of the study.
Arm/Group | APL + OBT
Number analyzed (Participants) | 0

23. Secondary Outcome: Plasma GW873140 400 mg BID PK Parameter of Maximum Observed Plasma Concentration (Cmax) During the Randomized Treatment Phase
Description: Cmax is defined as the first occurrence of the maximum observed plasma concentration determined directly from the raw concentration-time data. Blood samples for evaluation of GW873140 plasma PK was planned to be collected from all participants at Week 4, 12, and 24. Intensive PK sampling was planned to be conducted with the enrolled participants. All participants who were not part of the intensive PK group was planned to be part of the limited PK sample group. Participants were supposed to complete a diary card with the date and time of investigational product administration of the last dose prior to clinic visits on Weeks 4, 12, and 24.
Time Frame: as for outcome 22
Population: PK Population. Data were not collected for this outcome measure due to early termination of the study.
Arm/Group | APL + OBT
Number analyzed (Participants) | 0

24. Secondary Outcome: Plasma GW873140 400 mg BID PK Parameter of Time of Maximum Observed Plasma Concentration (Tmax) During the Randomized Treatment Phase
Description: Tmax is defined as the time at which Cmax is observed, determined directly from the raw concentration-time data. Blood samples for evaluation of GW873140 plasma PK was planned to be collected from all participants at Week 4, 12, and 24. Intensive PK sampling was planned to be conducted with the enrolled participants. All participants who were not part of the intensive PK group was planned to be part of the limited PK sample group. Participants were supposed to complete a diary card with the date and time of investigational product administration of the last dose prior to clinic visits on Weeks 4, 12, and 24.
Time Frame: as for outcome 22
Population: PK Population. Data were not collected for this outcome measure due to early termination of the study.
Arm/Group | APL + OBT
Number analyzed (Participants) | 0

25. Secondary Outcome: Plasma GW873140 400 mg BID PK Parameter of Concentration at End of Dosing Interval (Trough Concentration [Cτ]) During the Randomized Treatment Phase
Description: Blood samples for evaluation of GW873140 plasma PK was planned to be collected from all participants at Week 4, 12, and 24. Intensive PK sampling was planned to be conducted with the enrolled participants. All participants who were not part of the intensive PK group was planned to be part of the limited PK sample group. Participants were supposed to complete a diary card with the date and time of investigational product administration of the last dose prior to clinic visits on Weeks 4, 12, and 24.
Time Frame: as for outcome 22
Population: PK Population. Data were not collected for this outcome measure due to early termination of the study.
Arm/Group | APL + OBT
Number analyzed (Participants) | 0

26. Secondary Outcome: Investigational Product Adherence Measured by Pill Counts
Description: Adherence to investigational product was planned to be evaluated using pill counts of unused investigational product (blinded GW873140 or placebo, open-label GW873140 for open label phase). This assessment was planned to be conducted at each time the participant received a new (refill) supply of study medication.
Time Frame: Up to Week 48 of Randomized Treatment phase and up to Switch + 24 Weeks of the Open Labeled phase
Population: ITT Population. Data for this outcome measure were not collected due to early termination of the study.
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Number of Participants Who Were Bothered by Each of Several Specific Symptoms Evaluated Using the HIV Symptom Index Questionnaire During the Randomized Treatment Phase
Description: The HIV Symptom Index Questionnaire was planned to be used to evaluate how bothersome certain symptoms were during the conduct of this clinical study. The participant self-report instrument had 20 items, each of which asked about a specific symptom or group of related symptoms that participants might have had during the past 4 weeks and the degree to which the participant is bothered by the symptom. The symptom index comprised 32 common and HIV-specific symptoms scored in terms of presence/absence (1, 0) and severity on a 4-point scale (0 = not at all to 3 =quite a bit). Higher score represented greater severity of symptoms.
Time Frame: Upto Week 48
Population: ITT Population. Data for this outcome measure were not collected due to early termination of the study.
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 0 | 0

28. Secondary Outcome: Number of Participants With the Impact on Health Related Quality of Life Measured by Euro Quality of Life (Qol) Questionnaire During the Randomized Treatment Phase
Description: The EuroQol is a standardized instrument for use as a measure of health related quality of life. It consists of two pages comprising the EuroQoL 5 Dimension 5 level (EQ-5D5) descriptive system and the EQ visual analogue scale (VAS). The EQ-5D5 comprises of five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety). Each dimension comprises five levels of response (no problems, mild problems, moderate problems, moderate to extreme problems, and extreme problems). The EQ VAS records the respondents self-rated health status on a vertical graduated (0 to 100) VAS. Higher score represented greater severity of diseases.
Time Frame: Up to Week 48
Population: ITT Population. Data for this outcome measure were not collected due to early termination of the study.
Arm/Group | APL + OBT | Placebo + OBT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE's were collected up to Follow-up (Week 52)
Description: ITT Population was used.
Arm/Group | APL + OBT | Placebo + OBT
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 11/13 | 5/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | APL + OBT (N=13) | Placebo + OBT (N=11)
Diarrhoea (Gastrointestinal disorders) | 7 | 2
Nausea (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Rectal lesion (Gastrointestinal disorders) | 1 | 0
Stomach discomfort (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 0
Injection site pain (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Acarodermatitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Tinea cruris (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 0 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Study was early terminated prior to the completion of enrollment due to treatment-emergent hepatotoxicity that occurred among some participants receiving APL.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.